CLINICAL TRIAL: NCT04850989
Title: Efficacy of Using Real-Life Footage in Virtual Reality Exposure Therapy for Social Anxiety Disorder
Brief Title: Efficacy of Virtual Reality Exposure Therapy Scripts for Social Phobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Limbix Health, Inc. (Industry)
Responsible Party: Principal Investigator, Michelle G. Newman, Professor of Psychology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00010344
Record Dates: First submitted 2021-04-09; First posted 2021-04-20 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Social Anxiety Disorder
Keywords: Virtual reality; Exposure therapy; Self-help
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Intervention Model Description: Refer to published trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Virtual reality exposure therapy (Experimental): Participants were allowed to choose one of two themes. For both themes, each scene was developed to be more anxiety-provoking as the VRE progressed. Greater anxiety-inducing scenes had interviewers and other actors who displayed less compassionate, friendly, humorous, and pleasant verbal and non-verbal behaviors and demeanors to elicit elevated anxiety (Carless & Imber, 2007). Also, a virtual therapist was embedded within the VRE. It functioned to coach the participant through each distinct scene by orienting and prompting them to the exposure therapy task(s), continually conveying core principles of exposure therapy, and repeating the instructions if the participant was not responsive within five seconds. Each scene started with a paused video, during which participants were oriented by the virtual therapist to the context.
  Interventions: Device: Pico Goblin VR headset
- Waiting list (No Intervention): Participants started treatment 2-4 weeks post-randomization.

INTERVENTIONS:
Device: Pico Goblin VR headset — We worked with Limbix to tailor content on a Pico Goblin VR headset by creating two exposure therapy themes (general social skills training/dinner party or job interview) based on CBT principles and literature. The Pico Goblin VR headset projected a 5.5-inch diagonal screen size (depth: 139.7 mm; height: 122mm; width: 68mm) with 2560 x 1440-pixel resolution, 3 degrees of freedom, 92° field of view, a refresh rate of 70Hz, and 54-71mm interpupillary distance (Kyoto, 2017). It was chosen because displays of the pre-recorded VRE videos could be smoothly operated wirelessly with a tablet that showed the selected scenes in real-time. Further, the headset could be conveniently switched on and off, and dovetailed the participant's head motion. These scenes were filmed with a 360° stereoscopic camera, each lasting between 1.5 to 10 min.
  Arms: Virtual reality exposure therapy

SUMMARY:
The purpose of this study is to test the efficacy virtual reality videos to facilitate exposure therapy in social anxiety disorder (SAD). The exposure therapy videos are the focus of this experiment. Essentially, we are testing the efficacy of the Virtual Reality Exposure Therapy (VRET) scripts (i.e., virtual scenarios, people, and interactions that we expose socially anxious people to). To this end, the goal of the current study is to help people with social anxiety overcome their phobias. Individuals who experience a difficult time building social relationships, accomplishing everyday tasks, or pursuing job interviews can practice those same behaviors in a controlled environment. Specifically, we aim to test the following hypotheses: (1) Virtual reality exposure therapy intervention (vs. waitlist control condition) is effective for treating SAD symptoms. (2) Participants who received the VRET will experience maintenance of treatment gains following 3-month and 6-month post-termination of treatment. (3) Users of the virtual reality exposure therapy will demonstrate high amounts of acceptability of the treatment.

DETAILED DESCRIPTION:
Social anxiety disorder (SAD) is a widespread mental health problem (Kessler et al., 2012), marked by persistent and intense fear and avoidance of interpersonal situations that may be evaluative (American Psychiatric Association, 2013). SAD is acknowledged to be a complex condition that can be chronic or unremitting (Vriends, Bolt, & Kunz, 2014). Relatedly, persons with SAD tend to display compromised work or school functioning, relationship satisfaction, and quality of life (Teo, Lerrigo, & Rogers, 2013), as well as increased comorbid physical and mental health problems (Jacobson & Newman, 2017; Schmidt, Keough, Hunter, & Funk, 2008). Therefore, designing and delivering efficacious treatments for SAD is important.

Novel state-of-the-art psychotherapies for SAD have been developed. These include cognitive bias modification approaches (e.g., video feedback, imagery rescripting), cognitive behavioral therapies (CBT; e.g., social skills training, behavioral experiments), internet CBT, and neuroenhancers (e.g., D-cycloserine, yohimbine) (Stangier, 2016). Exposure therapy is a well-established, gold-standard efficacious specific CBT component for SAD (Otte, 2011). Such exposure therapy is grounded in emotional processing theory (Foa & Kozak, 1986), which proposes that fear memories can be interpreted as structures that store data concerning events, responses, and meaning propositions. By activating and altering fear structures, it is thought that exposure therapy can ease emotional processing through gradual and recurrent experiences of distress-evoking yet potentially rewarding and physically safe social interactions (Zalta & Foa, 2012). Specifically, exposure therapy is supposed to activate the fear structure by involving the person with SAD in various anxiety-provoking social situations to adjust the fear structure via habituation (reduced fear after repeated encounters of phobic situations) and extinction (unlearning of acquired fear connections; Furlong, Richardson, & McNally, 2016). On the other hand, it is plausible that even if within- or between-session habituation did not occur, extinction learning might be achieved via practicing greater fear tolerance in diverse anxiety-evoking social situations (cf. inhibitory learning theory; Craske et al., 2008). Relatedly, the cognitive model of SAD (Leigh & Clark, 2018) posits that exposure therapy works by improving psychological flexibility and other (vs. self-) focused attention as well as eliminating safety behaviors and threat hypervigilance, during anxiety-inducing social events.

Exposure therapy can be carried out in vivo (directly engaging with fear-evoking situations) or in vitro or imaginarily (continually visualizing exposure scenarios). However, in vivo exposure therapy can be time-consuming, costly, and how events unfold during exposure can neither be predicted nor controlled. Also, in vitro exposure therapy can be difficult and ineffective for highly-avoidant persons who lack the ability to envision specific scenes in clear detail and to stay in the imagined anxiety-inducing scenarios long enough for the imaginal exposure therapy to be effective (Hembree & Cahill, 2007; Vrielynck & Philippot, 2009). Thus, virtual reality exposure therapy (VRE) has been designed as a means for persons with SAD to privately immerse in myriad computer-generated fear-provoking social situations that mimic the natural environment (Anderson, Rothbaum, & Hodges, 2003). VRE offers latitude for the psychologist to construct exposure situations, receives more acceptance from patients, provides greater privacy, and has lower dropout rates than in vivo exposure therapy (Garcia-Palacios, Botella, Hoffman, & Fabregat, 2007; Krijn, Emmelkamp, Olafsson, & Biemond, 2004). Further, most clinicians have viewed VRE favorably (Lindner et al., 2019a).

To date, seven randomized controlled trials (RCTs) have examined the impact of therapist-directed VRE compared to waiting list (WL) for SAD. An early study showed that four therapist-facilitated 12-to-15-minute sessions of VRE (vs. WL) efficaciously reduced public speaking phobia for highly anxious college students from baseline to post-treatment (Harris, Kemmerling, & North, 2002); despite this reduction, VRE was not superior to WL in lowering SAD symptoms. Another four-session VRE (vs. WL) that instructed participants to repeatedly read a children's book to a virtual audience observed reductions in public speaking fear across time (Lister, Piercey, & Joordens, 2010); however, there were no changes on trait anxiety or social phobia symptoms. Relatedly, compared to WL, a therapist-guided, 12-session, VRE with various fear-inducing interpersonal situations led to decrements in SAD fear and avoidance severity, as well as public speaking phobia, among young adult females with public speaking anxiety (Wallach, Safir, & Bar-Zvi, 2011). Further, some sustained treatment gains at 1-year follow-up were observed (Safir, Wallach, & Bar-Zvi, 2012); however, high-anxious participants were not assessed for diagnoses of SAD in that study. In a similar nine-session, therapist-directed VRE (vs. WL) RCT for public speaking anxiety that additionally recruited patients with SAD and assigned between-session homework, large effect sizes for treatment efficacy were observed from baseline to 1-year follow-up (Anderson et al., 2013); nonetheless, findings may not extend beyond persons who had expressed public speaking fear as their main problem. Relatedly, VRE (vs. WL) was more effective in reducing avoidance and unhelpful beliefs as well as increasing speech duration in persons with SAD whose interpersonal fears extended to numerous contexts (Kampmann et al., 2016). Additionally, cognitive behavioral therapy (CBT) plus VRE (vs. WL) targeting multiple social fears was more effective at decreasing SAD severity (Bouchard et al., 2017); however, as it examined VRE blended with CBT, the efficacy of self-guided VRE as a stand-alone treatment could not be deduced.

Most of the VRE conducted so far has been therapist-led but attempts toward decreasing therapist participation have recently been underway. For example, one-session of minimally-therapist-assisted VRE (vs. in vivo exposure therapy) produced comparable reduction in behavioral avoidance frequency and fear severity in spider phobic individuals (Miloff et al., 2019). Likewise, completely self-guided, smartphone app-delivered VRE (vs. WL) resulted in large decreases in fear of heights for persons with acrophobia (Donker et al., 2019), with strong engagement across unique exposure scenarios that evoked varying degrees of fear (Donker, van Klaveren, Cornelisz, Kok, & van Gelder, 2020). In addition, the large effect of a relatively inexpensive, one-session, self-directed, Google Cardboard headset-delivered VRE for public speaking phobia did not differ significantly from a therapist-guided treatment (Lindner et al., 2019b). Such efforts are important to test further as VR can enhance the delivery of self-help exposure therapy to persons with SAD by decreasing costs and increasing access when trained therapists are not available. For example, it could decrease costs if used as part of a stepped care model. All patients within a health management organization (HMO) who could benefit from VRE, could first be assigned to complete self-guided VRE within a clinic. The clinic might contain multiple VRE equipped rooms and overseen by one minimum wage paid staff person who serves as a technician troubleshooting any mechanical faults with the equipment. If this was not sufficient to lead to remission the patient would then be provided more intensive in-person CBT with a well-trained and qualified CBT practitioner (Boeldt, McMahon, McFaul, & Greenleaf, 2019; Newman, Szkodny, Llera, & Przeworski, 2011). Alternatively self-help VRE equipment could be rented and/or purchased and used at home as the price of VRE devices has been declining across time (Bun, Gorski, Grajewski, Wichniarek, & Zawadzki, 2017).

Accordingly, building on prior work, we aimed to examine the efficacy of self-guided VRE for persons with SAD. There are several innovative aspects of the VRE used in the current study. First, our VRE had a virtual therapist built into it who auditorily guided participants through the exposure exercises and who conveyed CBT principles (see online supplementary material (OSM) for therapist script examples). We are aware of only one prior self-help VRE controlled trial that included a virtual therapist and this was for a treatment for acrophobia (Donker et al., 2019). The use of the virtual therapist also adds to prior work on non-self-help VREs (Anderson et al., 2013; Bouchard et al., 2017; Harris et al., 2002). Relatedly, the VRE included a built-in system to deliver and record subjective units of distress (SUDS) ratings. Further, it detected if the participant talked in response to the lifelike human character (professional actors were hired to play these roles) and the characters would wait until the participant provided verbal output before continuing the preprogrammed interaction). The current study also augments prior self-guided VRE controlled trials that did not contain cutting-edge, omnidirectional (360°), and dynamic video technology driven by machine learning optimization algorithms, biometrics, and programming rules (Lindner et al., 2019b; Lister et al., 2010). Also, to our knowledge, no other self-help controlled VRE study for SAD conducted exposure to bidirectional social interactions (Lindner et al., 2019b; Lister et al., 2010). Moreover, our study provided between-session exposure homework exercises to consolidate learning; a procedure mirroring face-to-face CBT but not conducted by any other self-help VRE study to date and omitted by more than half of the prior non-self-help studies on VRE for anxiety disorders thus far (refer to meta-analysis by Benbow & Anderson, 2019).

We hypothesized that from baseline to post-treatment, self-guided VRE would result in substantially greater decrease in primary outcomes (SAD severity and job interview anxiety) when compared to WL. Further, we hypothesized that VRE (vs. WL) would lead to larger reductions in secondary outcomes, namely trait worry and depression symptom severity. In addition, we anticipated that pre-post-treatment gains would be maintained across 3-month follow-up (3MFU) and 6-month follow-up (6MFU) periods. Lastly, we conducted exploratory analyses to examine whether there would be enhancement in presence (i.e., sense of virtual world mimicking real-life scenarios) and reduction in cybersickness across VRE sessions.

ELIGIBILITY:
Inclusion Criteria:

* Presence of Social Anxiety Disorder based on the Social Phobia Diagnostic Questionnaire self-report or Mini International Neuropsychiatric Interview
* Current student at the Pennsylvania State University or a community-dwelling adult who expressed interest to participate through the PSU StudyFinder portal
* Expressed interest to seek treatment
* Currently not receiving treatment from a mental health professional
* Able to provide consent
* Proficient in English

Exclusion Criteria:

* Below age 18
* Failure to meet any of above inclusion criteria
* Presence of suicidality, mania, psychosis, or substance use disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle G. Newman, Ph.D., Principal Investigator — The Pennsylvania State University
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Virtual Reality Exposure Therapy (VRE): We collaborated with a VR company, Limbix (https://www.limbix.com; now associated with BehaVR), that develops and provides VR-based mental health treatments (Paul, Bullock, & Bailenson, 2020; Summers, Schwartzberg, & Wilhelm, 2021). Specifically, we worked with Limbix to script the VR actors' verbal and non-verbal behaviors, virtual therapist's instructions, task prompts, and treatment rationale content in all scenes shown on a Pico Goblin VR headset. Two exposure therapy themes were created (informal dinner party or formal job interview) based on CBT principles and the literature. The headset displayed a 5.5-inch diagonal screen size (depth: 139.7 mm; height: 122mm; width: 68mm) with 2560 x 1440-pixel resolution, 3 degrees of freedom, 92° field of view, a refresh rate of 70Hz, and 54-71mm interpupillary distance (Kyoto, 2017). The VRE also contained cutting-edge 360° stereoscopic views allowing for an omnidirectional range of visual perspective as participants could look in all directions within the virtual environment. It also contained dynamic video technology driven by machine learning optimization algorithms, biometrics, and programming rules (Lindner et al., 2019b; Lister et al., 2010). With respect to biometrics, it had the ability to detect voice output (e.g., a person not speaking served as a precondition to virtual therapist prompts to speak with the avatar).
- Waitlist: Participants on the waitlist received the VRE treatment 4 weeks after the initial study visit.
Period: Overall Study
Arm/Group | Virtual Reality Exposure Therapy (VRE) | Waitlist
Started | 26 | 18
Completed | 21 | 14
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Virtual Reality Exposure Therapy: Self-Guided Virtual Reality Exposure Therapy
- Waitlist Control: Participants received the Virtual Reality Exposure Therapy after 2 weeks from the initial study visit.
- Total: Total of all reporting groups
Arm/Group | Virtual Reality Exposure Therapy | Waitlist Control | Total
Number analyzed (Participants) | 26 | 18 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.35 (8.63) | 23.22 (10.51) | 23.30 (9.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 34
  Male | 7 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Non-White | 13 | 8 | 21
  Race: White Caucasian | 13 | 10 | 23
Social Phobia Diagnostic Questionnaire (SPDQ) [Mean (Standard Deviation); unit: units on a scale] — The 25-item Diagnostic and Statistical Manual-Fourth Edition-Text Revised (DSM-IV-TR)-aligned Social Phobia Diagnostic Questionnaire (SPDQ; Newman, Kachin, Zuellig, Constantino, & Cashman-McGrath, 2003) was used to assess degree of fear and avoidance related to diverse social situations. Possible total scores (summed across all items) range from 0 to 27. A higher total score means a worse outcome.
  units on a scale | 19.12 (3.50) | 16.99 (4.42) | 18.06 (3.96)
Social Interaction Anxiety Scale (SIAS) [Mean (Standard Deviation); unit: units on a scale] — The 20-item Social Interaction Anxiety Scale (SIAS; Mattick & Clarke, 1998) was also used to assess SAD symptom severity. Participants rated on a 5-point Likert scale (0 = not at all characteristic or true of me to 4 = extremely characteristic or true of me) their degree of anxiety regarding social interactions. Possible total scores (summed across all items) range from 0 to 80. A higher total score means a worse outcome.
  units on a scale | 53.48 (9.53) | 46.45 (14.54) | 49.97 (12.04)
Measure of Anxiety in Selection Interviews (MASI) [Mean (Standard Deviation); unit: units on a scale] — The 30-item Measure of Anxiety in Selection Interviews (MASI; McCarthy & Goffin, 2004) was used to assess job interview anxiety severity. Respondents endorsed on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree) the degree to which they experienced anxiety surrounding appearance, behavioral, communication, performance, and social aspects of interviewing (e.g., "I become very uptight about having to interact with a job inter- viewer socially"). Possible total scores (summed across all items) range from 30 to 150. Higher scores denoted greater job interview anxiety.
  units on a scale | 74.87 (15.80) | 70.46 (16.27) | 72.67 (16.04)
Penn State Worry Questionnaire (PSWQ) [Mean (Standard Deviation); unit: units on a scale] — The 16-item Penn State Worry Questionnaire (PSWQ; Meyer, Miller, Metzger, & Borkovec, 1990) was utilized to measure trait worry. Participants rated the extent to which they tended to worry excessively on a 5-point Likert scale (1 = not typical at all to 5 = very typical). Possible total scores (summed across all items) range from 16 to 80. Higher scores denoted stronger trait worry.
  units on a scale | 67.60 (6.92) | 60.19 (7.81) | 63.90 (7.37)
Patient Health Questionnaire (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — The 9-item Patient Health Questionnaire (PHQ-9; Kroenke, Spitzer, & Williams, 2001) was used to assess extent of depression symptom severity. Respondents rated the frequency with which they encountered depression symptoms in the past 2 weeks on a 4-point Likert scale (0 = Not at all to 3 = Nearly every day). Possible total scores (summed across all items) range from 0 to 27. Higher scores denoted stronger depression symptom severity.
  units on a scale | 13.20 (5.80) | 11.20 (6.01) | 12.20 (5.91)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Social Phobia Diagnostic Questionnaire (SPDQ) at Post-treatment
Description: The 25-item Diagnostic and Statistical Manual-Fourth Edition-Text Revised (DSM-IV-TR)-aligned Social Phobia Diagnostic Questionnaire (SPDQ; Newman, Kachin, Zuellig, Constantino, & Cashman-McGrath, 2003) is a self-report instrument designed to assess the degree of fear and avoidance associated with various social situations. Each item evaluates the severity of fear and the frequency of avoidance on a 5-point Likert scale, where 0 indicates "no fear" or "never avoid," and 4 signifies "very severe fear" or "always avoid" . The total score is derived by summing the responses across all items, yielding a range from 0 to 27, with higher scores reflecting greater social anxiety symptoms . In clinical trials, change scores are calculated by subtracting post-treatment scores from baseline scores, resulting in a possible range from -27 to 27; higher (less negative) change scores indicate better outcomes, signifying a reduction in social anxiety symptoms.
Time Frame: Baseline and post-treatment, on average 2 weeks
Population: Intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Virtual Reality Exposure Therapy: Participants engaged with the virtual reality exposure therapy designed to last four sessions or more.
- Waitlist Control: Participants on the waitlist received the virtual reality exposure therapy four weeks post-randomization.
Arm/Group | Virtual Reality Exposure Therapy | Waitlist Control
Number analyzed (Participants) | 26 | 18
score on a scale | -9.60 (0.01) | -4.46 (0.50)
Statistical Analysis 1: Comparison: Virtual Reality Exposure Therapy vs Waitlist Control; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Net) = -5.14, Standard Deviation 0.49

2. Primary Outcome: Change From Baseline in the Social Interaction Anxiety Scale (SIAS) at Post-treatment
Description: The 20-item Social Interaction Anxiety Scale (SIAS; Mattick & Clarke, 1998) is a self-report instrument designed to assess the severity of social anxiety disorder (SAD) symptoms, particularly focusing on distress experienced during social interactions. Each item is rated on a 5-point Likert scale ranging from 0 ("not at all characteristic or true of me") to 4 ("extremely characteristic or true of me"), yielding a total score between 0 and 80. Notably, items 5, 9, and 11 are reverse-scored. Higher total scores indicate greater levels of social interaction anxiety. Clinically, a total score of 36 or above suggests probable social anxiety disorder, while a score of 43 or higher indicates SAD. Change scores are calculated by subtracting the post-treatment score from the pre-treatment score, resulting in a possible range from -80 to 80. Negative change scores (i.e., a decrease in total SIAS score) reflect a reduction in social anxiety symptoms, thus indicating better outcomes.
Time Frame: Baseline and post-treatment, on average 2 weeks
Population: Intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Exposure Therapy | Waitlist Control
Number analyzed (Participants) | 26 | 18
score on a scale | -28.19 (0.03) | -16.65 (1.26)
Statistical Analysis 1: Comparison: Virtual Reality Exposure Therapy vs Waitlist Control; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Net) = -11.54, Standard Deviation -1.23

3. Secondary Outcome: Change From Baseline in the Measure of Anxiety in Selection Interviews (MASI) at Post-treatment
Description: The 30-item Measure of Anxiety in Selection Interviews (MASI; McCarthy & Goffin, 2004) is a self-report designed to assess the severity of job interview anxiety across five dimensions: communication anxiety, appearance anxiety, social anxiety, performance anxiety, and behavioral anxiety. Each item is rated on a 5-point Likert scale ranging from 1 ("strongly disagree") to 5 ("strongly agree"), resulting in a total score range from 30 to 150, with higher scores indicating greater levels of interview anxiety. Change scores are calculated by subtracting the post-treatment score from the pre-treatment score, yielding a possible range from -120 to 120; larger negative change scores reflect a reduction in interview anxiety symptoms, thus indicating better outcomes.
Time Frame: Baseline and post-treatment, on average 2 weeks
Population: Intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Exposure Therapy | Waitlist Control
Number analyzed (Participants) | 26 | 18
score on a scale | -36.52 (1.08) | -22.57 (6.21)
Statistical Analysis 1: Comparison: Virtual Reality Exposure Therapy vs Waitlist Control; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Net) = -8.08, Standard Deviation 1.91

4. Secondary Outcome: Change From Baseline in the Penn State Worry Questionnaire (PSWQ) at Post-treatment
Description: The 16-item Penn State Worry Questionnaire (PSWQ; Meyer, Miller, Metzger, & Borkovec, 1990) is a self-report instrument designed to assess the trait of pathological worry, a core feature of generalized anxiety disorder (GAD). Each item is rated on a 5-point Likert scale ranging from 1 ("not at all typical of me") to 5 ("very typical of me"), yielding total scores between 16 and 80. Higher scores indicate greater severity of worry. The PSWQ includes 11 items that directly assess worry and 5 reverse-scored items that measure the absence of worry, which must be recoded before computing the total score . In clinical trials, change scores are calculated by subtracting the post-treatment score from the pre-treatment score, resulting in a possible range from -64 to 64; larger negative change scores reflect a reduction in worry symptoms, thus indicating better outcomes.
Time Frame: Baseline and post-treatment, on average 2 weeks
Population: Intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Exposure Therapy | Waitlist Control
Number analyzed (Participants) | 26 | 18
score on a scale | -21.18 (1.81) | -13.10 (0.10)
Statistical Analysis 1: Comparison: Virtual Reality Exposure Therapy vs Waitlist Control; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Net) = -8.08, Standard Deviation 1.91

5. Secondary Outcome: Change From Baseline in the Patient Health Questionnaire (PHQ-9) at Post-treatment
Description: The 9-item Patient Health Questionnaire (PHQ-9; Kroenke, Spitzer, & Williams, 2001) is a self-administered instrument designed to assess the severity of depressive symptoms over the past two weeks, based on the diagnostic criteria outlined in the DSM-IV. Each item is rated on a 4-point Likert scale ranging from 0 ("Not at all") to 3 ("Nearly every day"), resulting in a total score that can range from 0 to 27. Higher scores correspond to more severe depressive symptoms, with established cutpoints indicating depression severity as follows: 0-4 (none or minimal), 5-9 (mild), 10-14 (moderate), 15-19 (moderately severe), and 20-27 (severe) . In clinical trials, change scores are calculated by subtracting the post-treatment score from the pre-treatment score, yielding a possible range from -27 to 27; positive change scores reflect a reduction in depressive symptoms, indicating better outcomes.
Time Frame: Baseline and post-treatment, on average 2 weeks
Population: Intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Exposure Therapy | Waitlist Control
Number analyzed (Participants) | 26 | 18
score on a scale | -6.74 (2.69) | -3.26 (2.41)
Statistical Analysis 1: Comparison: Virtual Reality Exposure Therapy vs Waitlist Control; Test type: Superiority; p > 0.05, Mixed Models Analysis; Mean Difference (Net) = -3.48, Standard Deviation 0.28

ADVERSE EVENTS:
Time Frame: Adverse events were neither assessed nor monitored during this trial.
Description: Adverse events were neither assessed nor monitored during this trial.
Groups:
- Waiting List: Participants on the waitlist received the virtual reality exposure therapy four weeks post-randomization.
Arm/Group | Virtual Reality Exposure Therapy | Waiting List
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT04850989/Prot_SAP_ICF_002.pdf